CLINICAL TRIAL: NCT06233214
Title: The Effect of the Vein Imaging Device Used in Peripheral Intravenous Catheter Application on the Success of the Procedure in Patients Coming to the Pediatric Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: vein imaging
Record Dates: First submitted 2023-12-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Intravenous Catheter
Keywords: pediatrics; peripheral intravenous catheter application; vein imaging device

STUDY DESIGN:
Intervention Model Description: PIC placement attempt will be performed with the help of a vein imaging device in the study/experiment group, and with the traditional application method without device support in the control group.
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vein imaging device (Experimental): During the PIC application attempt, the parents of the children in the experimental group will be ensured to be with their children throughout the procedure.
  PIC placement attempt will be performed on the experimental group with the help of a vein imaging device.
  Interventions: Device: vein imaging device
- control group (No Intervention): PIC placement attempt will be performed in the control group using the traditional application method without device support.

INTERVENTIONS:
Device: vein imaging device — During the PIC application attempt, the parents of the children in the experimental group will be ensured to be with their children throughout the procedure.
  PIC placement attempt will be performed on the experimental group with the help of a vein imaging device.
  Arms: vein imaging device

SUMMARY:
Peripheral Intravenous Catheter (PIC) application in pediatric wards of hospitals; It is used in the administration of drugs that require diarrhea, vomiting, dehydration or high serum concentration, resistant infections, parenteral treatments, continuous bolus analgesic needs and emergency treatment situations. Although PIC is a frequently used practice, especially in pediatric emergency departments, it is seen as a difficult approach for healthcare professionals. PIC applications may be more difficult in pediatric patients due to their small vascular structures, the fact that the vessels are surrounded by subcutaneous tissue, and lack of communication. Every child's venous anatomy is different. Therefore, selecting the appropriate vein by ensuring palpation and using appropriate tools before the procedure will reduce the pain and stress the child will experience. Biomedical tools are used to increase success in vascular interventions. Studies have shown that PIC procedure time is shorter in pediatric patients using vein imaging devices and the number of interventions is lower than the control group.

DETAILED DESCRIPTION:
Assistive devices may be needed to perform this procedure, which is quite painful and anxiety-inducing for children, all at once and in a short time. In this regard, there is no device support for PIC application for pediatric patients at Manisa Celal Bayar University Hafsa Sultan Hospital. The investigators predict that by introducing the vein imaging device to the Pediatric Emergency Department of our hospital, the success rate of PIC application will increase and the number of interventions will decrease by enabling the vein to be visualized and selected in pediatric patients. Due to these processes experienced by pediatric patients, the aim of our research is to examine the effect of the vein imaging device used during peripheral intravenous catheter application on the success of the procedure in pediatric patients. Method: The population of the research will consist of pediatric patients between the ages of 6-12 who applied to the Pediatric Emergency Department of Manisa Celal Bayar University, Hafsa Sultan Hospital. The adequacy of the sample size in the study "G. Calculated using the "Power-3.1.9.2" program. In the power analysis performed for the sample and power calculation of the experimental study, 30 pediatric patients were determined for each group at the p = 0.05 level, 80% representative power of the population and 95% confidence interval. However, considering the missing data, it was planned to conduct a study with 35 children for the experimental and control groups. Randomization was performed using the random numbers table obtained from the computer program (https://www.randomizer.org/).

Research data will be collected at Manisa Celal Bayar University Hafsa Sultan Hospital Pediatric Emergency Service. The research was planned as an experimental (n: 35) and control (n: 35) group.

In collecting data;

* Informed Volunteer Consent Form (Appendix I).
* Interview and Observation Form (Annex II).
* Challenging Intravenous Intervention Score for Children (Appendix III).
* ACCUVEIN AV 500 vein imaging device (Annex IV)
* Peripheral cannula (Yellow color No. 24 G or Blue color No. 22 G) (Annex V): will be used.

Data collection phase; Pediatric patients and their families who come to the pediatric emergency department will be informed about the vein imaging device to be used in the research and how the research will be conducted. Their consent will be taken. PIK placement attempt will be performed with the help of a vein imaging device in the experimental group, and with the traditional application method without device support in the control group. PIC placement in both groups will be performed by a specialist nurse working in the pediatric emergency department, who has 5 years of experience in caring for pediatric patients and performing IV interventions. In order to avoid differences in practice, the procedure for establishing peripheral vascular access for all children will be provided by the same nurse. In both groups, all PIK procedures will be performed with the same catheter number (24-G yellow or 22-G blue) and the same brand catheter (Braun) to avoid differences. Another pediatric emergency nurse who has been working in the pediatric emergency department for at least 2 years, independent of the research, will also act as an observer. When evaluating the duration of the PIK placement attempt; Before the child's vein is searched, the stopwatch will be turned on as soon as the tourniquet is tied and the time will be stopped when the patency of the vascular access is ensured (from the time the tourniquet is tied until the physiological saline is given). If the vascular access fails in the first attempt, a new vein will be searched and time will be kept until the procedure is successful. Once vascular access is established, the time will be stopped and the procedure time will be recorded. The observing nurse will evaluate the "Interview and Observation Form" and the "Difficult Intravenous Intervention Score for Children".

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 6-12,
* The child is receiving treatment through peripheral vascular access,
* Parent and child agree to participate in the research,
* PIK placement is done by the same nurse,
* PIK placement should be performed with the same catheter number (24-G or 22-G) and brand.

Exclusion Criteria:

Children falling outside the inclusion criteria will be included in the exclusion criteria.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Interview and Observation Form | it will take approximately 5 minutes to fill out the form.
  This form consists of 13 items developed based on the available literature. The first five items question demographic characteristics, and the others question the success of the procedure regarding the number of attempts and their duration.

SECONDARY OUTCOMES:
Difficult Intravenous Access Score | it will take approximately 1 minutes to fill out the form.
  It was developed by Yen et al. The DIVA score with 4 parameters (visibility, palpability, age, and prematurity history) was found to be valid and reliable for Turkish children. The vascular access is assessed as difficult with a 50% failure rate if the total score is 4 and above.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Karaarslan, Study Director — Manisa Celal Bayar University
Locations (1):
- Manisa Hafsa Sultan Hospital, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No